CLINICAL TRIAL: NCT03314545
Title: Clinical Evaluation of Laminate Veneers With Coronal Post Versus Post and Core Foundation Restoration With Single Crown for Restoration of Endodontically Treated Anterior Teeth (Randomized Controlled Trial) "In-vivo Study"
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Abdelrahman Elsadek, Assistant Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEBD-CU-2017-09-32
Record Dates: First submitted 2017-10-15; First posted 2017-10-19 (Actual); Last update posted 2017-10-19 (Actual); Status verified 2017-10

CONDITIONS: Teeth, Endodontically-Treated; Anterior Teeth
Keywords: endocrown; laminate veneer with coronal post; post and core; crown
MeSH Terms: conditions — Tooth, Nonvital | interventions — Crowns

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- laminate veneers with coronal posts (Other): anterior endodontically treated teeth restored with laminate veneers with coronal posts
  Interventions: Procedure: laminate veneer with coronal post
- post, core and crown (Other): anterior endodontically treated teeth restored with post, core and crown
  Interventions: Procedure: post,core and crown

INTERVENTIONS:
Procedure: laminate veneer with coronal post — laminate veneer with coronal post
  Other Names: anterior endocrown; endolam; endolaminate
  Arms: laminate veneers with coronal posts
Procedure: post,core and crown — post,core and crown
  Arms: post, core and crown

SUMMARY:
Clinical evaluation of Laminate veneers with coronal post versus post and core foundation restoration with single crown for restoration of endodontically treated anterior teeth (Randomized Controlled Trial) "In-vivo Study"

ELIGIBILITY:
Inclusion Criteria:

1. From 18-60 years old, should be able to read and sign the consent document.
2. Ability to tolerate the restorative procedures (physical and psychological).
3. Patients with anterior endodontically treated teeth indicated for coronal restoration:

   1. Good oral hygiene
   2. Minimum remaining coronal tooth height of 4 mm
   3. Normal functional occlusal stresses within physiological limits.
   4. Adequate crown/root ratio
   5. No signs and symptoms related to active periapical pathosis or endodontic failure.
4. With no active periodontal or pulpal problems.
5. Willing to return for follow-up visits.

Exclusion Criteria:

1. Teeth not fully erupted as in young patients.
2. Poor oral hygiene and lack of motivation
3. Vital teeth
4. Psychiatric problems or unrealistic expectations
5. Excessive parafunctional stresses and bad habits like nail biting. 11
6. The absence of sound enamel margins for the preparation
7. Abnormally small teeth or with structural defects in enamel. 12
8. Tooth mobility or inadequate crown/root ratio.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Estimated)
Dates: Start 2017-12 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Gross Fracture | one year
  : Alpha (A),Restoration is intact and fully retained. Bravo (B), Restoration is partially retained with some portion of the restoration still intact.
  Charlie (C), Restoration is completely missing.

SECONDARY OUTCOMES:
marginal integrity | one year
  Alpha (A), Visual inspection and explorer, the explorer does not catch when drawn across the surface of the restoration toward the tooth, or, if the explorer does not catch, there is no visible crevice along the periphery of the restoration. Bravo (B), Visual inspection and explorer, the explorer catches and there is visible evidence of a crevice, which the explorer penetrates, indicating that the edge of the restoration does not adapt closely to the tooth structure. The dentin and/or the base is not exposed, and the restoration is not mobile. Charlie (C), Explorer, the explorer penetrates crevice defect extended to the dentino-enamel junction.
marginal discoloration | one year
  Alpha (A) Visual inspection, There is no visual evidence of marginal discoloration different from the color of the restorative material and from the color of the adjacent tooth structure. Bravo (B), Visual inspection, There is visual evidence of marginal discoloration at the junction of the tooth structure and the restoration, but the discoloration has not penetrated along the restoration in a pulpal direction. Charlie (C), Visual inspection, there is visual evidence of marginal discoloration at the junction of the tooth structure and the restoration that has penetrated along the restoration in a pulpal direction.
color match | one year
  Alpha (A) Visual inspection The restoration appears to match the shade and translucency of adjacent tooth tissues. Bravo (B), Visual inspection, the restoration does not match the shade and translucency of adjacent tooth tissues, but the mismatch is within the normal range of tooth shades. (Within normal range: Similar to silicate cement restorations for which the dentist did not quite succeed in matching tooth color by his choice among available silicate cement shades.) Charlie (C), visual inspection , the restoration does not match the shade and translucency of the adjacent tooth structure, and the mismatch is outside the normal range of tooth shades and translucency.
caries | one year
  Alpha (A) Visual inspection, the restoration is a continuation of existing anatomic form adjacent to the restoration. Bravo (B), Visual inspection, there is visual evidence of dark deep discoloration adjacent to the restoration (but not directly associated with cavosurface margins).

IPD SHARING:
Plan to Share IPD: No